CLINICAL TRIAL: NCT06052059
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Program to Evaluate the Efficacy and Safety of MK-7240 in Participants With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Study to Evaluate Efficacy and Safety of Tulisokibart (MK-7240) in Participants With Moderately to Severely Active Ulcerative Colitis (MK-7240-001)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: PPD, Part of Thermo Fisher Scientific (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7240-001; PR200-301 (Other: PrometheusBio); jRCT2031230563 (Registry Identifier: jRCT); U1111-1296-0203 (Registry Identifier: UTN); U1111-1314-0050 (Registry Identifier: UTN); 2023-507473-17-00 (Registry Identifier: EU CT); 2024-518603-22-00 (Registry Identifier: EU CT)
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Ulcerative Colitis
Keywords: Inflammatory Bowel Disease
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Induction and maintenance treatments will be blinded. Reinduction will not be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (11):
- Study 1: High Dose Induction, High Dose Maintenance (Experimental): Participants receive high dose intravenous (IV) tulisokibart, followed by a high dose subcutaneous (SC) tulisokibart regimen.
  Interventions: Drug: IV Tulisokibart; Drug: SC Tulisokibart
- Study 1: High Dose Induction, Low Dose Maintenance (Experimental): Participants receive high dose IV tulisokibart, followed by a low dose SC tulisokibart regimen.
  Interventions: Drug: IV Tulisokibart; Drug: SC Tulisokibart; Drug: SC Placebo
- Study 1: Low Dose Induction, Low Dose Maintenance (Experimental): Participants receive low dose IV tulisokibart, followed by a low dose SC tulisokibart regimen.
  Interventions: Drug: IV Tulisokibart; Drug: SC Tulisokibart; Drug: SC Placebo
- Study 1: Placebo (Placebo Comparator): Participants receive IV placebo, followed by an SC placebo regimen.
  Interventions: Drug: IV Tulisokibart; Drug: IV Placebo; Drug: SC Placebo
- Study 1: High Dose Extension (Experimental): Participants receive a high dose SC tulisokibart regimen. Participants may be enrolled in this arm after completing participation in their original arm, if they meet protocol-specific prerequisites.
  Interventions: Drug: SC Tulisokibart
- Study 1: Low Dose Extension (Experimental): Participants receive a low dose SC tulisokibart and placebo regimen. Participants may be enrolled in this arm after completing participation in their original arm, if they meet protocol-specific prerequisites.
  Interventions: Drug: SC Tulisokibart; Drug: SC Placebo
- Study 2: High Dose Induction (Experimental): Participants receive high dose IV tulisokibart.
  Interventions: Drug: IV Tulisokibart
- Study 2: Low Dose Induction (Experimental): Participants receive low dose IV tulisokibart.
  Interventions: Drug: IV Tulisokibart
- Study 2: Placebo (Placebo Comparator): Participants receive IV placebo.
  Interventions: Drug: IV Tulisokibart; Drug: IV Placebo; Drug: SC Placebo
- Study 2: High Dose Extension (Experimental): Participants receive a high dose SC tulisokibart regimen. Participants may be enrolled in this arm only after completing participation in their original arm, if they meet protocol-specific prerequisites.
  Interventions: Drug: SC Tulisokibart
- Study 2: Low Dose Extension (Experimental): Participants receive a low dose SC tulisokibart regimen. Participants may be enrolled in this arm only after completing participation in their original arm, if they meet protocol-specific prerequisites.
  Interventions: Drug: SC Tulisokibart; Drug: SC Placebo

INTERVENTIONS:
Drug: IV Tulisokibart — Humanized monoclonal antibody that binds human tumor necrosis factor-like cytokine 1A (TL1A), administered intravenously
  Other Names: PRA023; MK-7240
  Arms: Study 1: High Dose Induction, High Dose Maintenance; Study 1: High Dose Induction, Low Dose Maintenance; Study 1: Low Dose Induction, Low Dose Maintenance; Study 1: Placebo; Study 2: High Dose Induction; Study 2: Low Dose Induction; Study 2: Placebo
Drug: IV Placebo — Placebo matching IV tulisokibart
  Arms: Study 1: Placebo; Study 2: Placebo
Drug: SC Tulisokibart — Humanized monoclonal antibody that binds human tumor necrosis factor-like cytokine 1A (TL1A), administered subcutaneously
  Other Names: PRA023; MK-7240
  Arms: Study 1: High Dose Extension; Study 1: High Dose Induction, High Dose Maintenance; Study 1: High Dose Induction, Low Dose Maintenance; Study 1: Low Dose Extension; Study 1: Low Dose Induction, Low Dose Maintenance; Study 2: High Dose Extension; Study 2: Low Dose Extension
Drug: SC Placebo — Placebo matching SC tulisokibart
  Arms: Study 1: High Dose Induction, Low Dose Maintenance; Study 1: Low Dose Extension; Study 1: Low Dose Induction, Low Dose Maintenance; Study 1: Placebo; Study 2: Low Dose Extension; Study 2: Placebo

SUMMARY:
The purpose of this protocol is to evaluate the efficacy of tulisokibart in participants with moderately to severely active ulcerative colitis. Study 1's primary hypotheses are that at least 1 tulisokibart dose level is superior to Placebo in the proportion of participants achieving clinical remission according to the Modified Mayo Score at Week 12, and that at least 1 tulisokibart dose level is superior to Placebo in the proportion of participants achieving clinical remission according to the Modified Mayo Score at week 52. Study 2's primary hypothesis is that at least 1 tulisokibart dose level is superior to Placebo in the proportion of participants achieving clinical remission according to the Modified Mayo Score at Week 12.

DETAILED DESCRIPTION:
The protocol consists of 2 studies. Study 1 includes induction and maintenance treatment, and Study 2 includes only induction treatment. Each study has its own hypotheses and outcome measures that will be assessed independently.

ELIGIBILITY:
Inclusion Criteria:

* Has had ulcerative colitis (UC) (from onset of symptoms) for at least 3 months before randomization
* Has moderately to severely active UC
* Weight ≥40 kg
* Satisfies at least 1 of the following criteria:

  * Has had an inadequate response or loss of response to 1 or more protocol-specified UC treatments
  * Protocol specified corticosteroid dependence
  * Has been intolerant to 1 or more protocol-specified UC treatments
* Is on treatment with any protocol-specified drugs during the study and meets drug stabilization requirements, as applicable
* Adolescent participants ≥16 and <18 years of age can participate if approved by the country or regulatory/health authority
* A participant assigned female sex at birth is eligible to participate if not pregnant or breastfeeding and Is not a participant of childbearing potential (POCBP); or is a POCBP and uses an acceptable contraceptive method, or is abstinent from penile-vaginal intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis), has a negative highly sensitive pregnancy test (urine or serum) as required by local regulations within 24 hours (for a urine test) or 72 hours (for a serum test) before the first dose of study intervention, medical history, menstrual history, and recent sexual activity has been reviewed by the investigator to decrease the risk for inclusion of a POCBP with an early undetected pregnancy

Exclusion Criteria:

* Has a diagnosis of Crohn's Disease (CD) or indeterminate colitis (inflammatory bowel disease (IBD)-undefined) or other types of colitis or enteritis that may confound efficacy assessment.
* Has a current diagnosis of fulminant colitis and/or toxic megacolon
* Has UC limited to the rectum (i.e, must have evidence of UC extending beyond the rectosigmoid junction, which is ~10 cm from the anal margin)
* Has a current or impending need for colostomy or ileostomy
* Has had a total proctocolectomy or partial colectomy
* Has received fecal microbial transplantation within 4 weeks before randomization
* Has had UC exacerbation requiring hospitalization within 2 weeks before screening
* Has prior or current evidence of definite colonic dysplasia except for low-grade dysplasia that has been completely removed
* Has any active or serious infections without resolution after adequate treatment
* Has had cytomegalovirus infection that resolved less than 4 weeks before screening
* Has a transplanted organ which requires continued immunosuppression
* Has a history of cancer (except fully treated non-melanoma skin cell cancers or cervical carcinoma in situ after complete surgical removal) within the last 5 years
* Is known to be infected with hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV)
* Has evidence of active tuberculosis (TB), latent TB not successfully treated (per local guidelines), or inadequately treated TB (for participants with history of TB)
* Has confirmed or suspected COVID-19
* Has a history of drug or alcohol abuse within 6 months prior to screening
* Has had major surgery within 3 months before screening or has a major surgery planned during the study
* Is currently receiving or is planning to receive total parenteral nutrition at any time during study treatment
* Has received UC-related antibiotics and has not been on stable doses for at least 14 days before randomization or has discontinued these medications within 14 days of randomization
* Requires treatment with a therapy that does not adhere to the protocol-specified guidance parameters
* Has received protocol-specified prohibited medications
* Has had prior exposure to tulisokibart or another anti-tumor necrosis factor-like cytokine 1A (TL1A) antibody

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1020 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Study 1: Percentage of Participants Achieving Clinical Remission Per Modified Mayo Score (MMS) at Week 12 | Week 12
  The Modified Mayo Score (MMS) is a composite score of ulcerative colitis (UC) disease activity on a scale of increasing severity from 0-9, calculated by summing three subscores: Endoscopic subscore (ES), scored on a scale of increasing severity from 0 (normal or inactive disease) to 3 (severe disease, such as spontaneous bleeding or ulceration); Stool frequency subscore (SFS), scored on a scale of increasing frequency from 0 (normal number of stools) to 3 (≥5 stools more than normal per day for the participant); and rectal bleeding subscore (RBS), scored on a scale of increasing severity from 0 (no blood seen) to 3 (blood alone passed). Clinical Remission is defined as an ES of 0 or 1, RBS of 0, and SFS of 0 or 1 and not greater than the baseline SFS.
Study 1: Percentage of Participants Achieving Clinical Remission Per MMS at Week 52 | Week 52
  The MMS is a composite score of UC disease activity on a scale of increasing severity from 0-9, calculated by summing three subscores: ES, scored on a scale of increasing severity from 0 (normal or inactive disease) to 3 (severe disease, such as spontaneous bleeding or ulceration); SFS, scored on a scale of increasing frequency from 0 (normal number of stools) to 3 (≥5 stools more than normal per day for the participant); and RBS, scored on a scale of increasing severity from 0 (no blood seen) to 3 (blood alone passed). Clinical Remission is defined as an ES of 0 or 1, RBS of 0, and SFS of 0 or 1 and not greater than the baseline SFS.
Study 2: Percentage of Participants Achieving Clinical Remission Per MMS at Week 12 | Week 12
  The MMS is a composite score of UC disease activity on a scale of increasing severity from 0-9, calculated by summing three subscores: ES, scored on a scale of increasing severity from 0 (normal or inactive disease) to 3 (severe disease, such as spontaneous bleeding or ulceration); SFS, scored on a scale of increasing frequency from 0 (normal number of stools) to 3 (≥5 stools more than normal per day for the participant); and RBS, scored on a scale of increasing severity from 0 (no blood seen) to 3 (blood alone passed). Clinical Remission is defined as an ES of 0 or 1, RBS of 0, and SFS of 0 or 1 and not greater than the baseline SFS.

SECONDARY OUTCOMES:
Study 1: Percentage of Participants With One or More Adverse Events (AEs) | Up to approximately 52 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants who experience an AE will be reported.
Study 1: Percentage of Participants Who Discontinued Study Intervention Due to an AE | Up to approximately 52 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinue study treatment due to an AE will be reported.
Study 1: Percentage of Participants Achieving Clinical Response Per Partial Modified Mayo Score (pMMS) at Week 2 | Week 2
  The partial Modified Mayo Score (pMMS) is a composite score of UC disease activity on a scale of increasing severity from 0-6, calculated by summing two subscores: SFS, scored from 0 (normal number of stools) to 3 (≥5 stools more than normal per day for the participant); RBS, scored from 0 (no blood seen) to 3 (blood alone passed). Clinical response is defined as pMMS reduction of 1 or more points and 30% or more, plus a reduction of 1 or more points in RBS or an absolute RBS of 0 or 1.
Study 1: Percentage of Participants With Endoscopic Improvement at Week 12 | Week 12
  Endoscopic improvement is defined as Mayo endoscopic subscore (ES) of 0 or 1. The ES measures UC severity based on endoscopy on a 0-3 scale of increasing severity.
Study 1: Percentage of Participants Achieving a Clinical Response Per MMS at Week 12 | Week 12
  The MMS is a composite score of UC disease activity on a scale of increasing severity from 0-9, calculated by summing three subscores: ES, scored on a scale of increasing severity from 0 (normal or inactive disease) to 3 (severe disease, such as spontaneous bleeding or ulceration); SFS, scored on a scale of increasing frequency from 0 (normal number of stools) to 3 (≥5 stools more than normal per day for the participant); and RBS, scored on a scale of increasing severity from 0 (no blood seen) to 3 (blood alone passed). Clinical response is defined as an MMS reduction of 2 or more points and 30% or more, plus a reduction of more than 1 point in RBS or an absolute RBS of 0 or 1.
Study 1: Percentage of Participants Achieving Histologic-Endoscopic Mucosal Improvement (HEMI) at Week 12 | Week 12
  HEMI is defined as a Geboes score of 3.1 or less and ES of 0 or 1. The Geboes score is a histologic grading system for inflammation in UC with scores ranging from 0 to 5.4, with higher scores indicating more severe inflammation. ES measures UC severity based on endoscopy, scored from 0 (normal or inactive disease) to 3 (severe disease, such as spontaneous bleeding or ulceration).
Study 1: Percentage of Participants Achieving Clinical Remission Per pMMS at Week 12 | Week 12
  pMMS is a composite score of UC disease activity on a scale of increasing severity from 0-6, calculated by summing two subscores: SFS, scored from 0 (normal number of stools) to 3 (≥5 stools more than normal per day for the participant); RBS, scored from 0 (no blood seen) to 3 (blood alone passed). Clinical remission per pMMS is defined as an RBS of 0 and SFS of ≤1.
Study 1: Percentage of Participants With Endoscopic Remission at Week 12 | Week 12
  ES measures UC severity based on endoscopy, scored from 0 (normal or inactive disease) to 3 (severe disease, such as spontaneous bleeding or ulceration). Endoscopic remission is defined as an ES of 0.
Study 1: Percentage of Participants Reporting No Bowel Urgency at Week 12 | Week 12
  Bowel urgency is measured using an NRS, which rates bowel urgency on a 0-11 scale of increasing severity. Resolution is defined as a score of 0 or 1 in participants who had a baseline score of 3 or more.
Study 1: Percentage of Participants Reporting No Abdominal Pain at Week 12 | Week 12
  Abdominal pain is measured on a 0-4 NRS of increasing pain severity. Absence of abdominal pain is defined as a rating of 0.
Study 1: Percentage of Participants Achieving Inflammatory Bowel Disease Questionnaire (IBDQ) Remission at Week 12 | Week 12
  The IBDQ measures health related quality of life in subjects with inflammatory bowel disease. It consists of 32 questions each with a graded response of 1 (worst) to 7 (best). The score ranges from 32 to 224. IBDQ remission is defined as a score of at least 170.
Study 1: Change from Baseline in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) Score at Week 12 | Baseline and Week 12
  The FACIT-Fatigue is a 13-item measure that assesses self-reported fatigue and its impact upon daily activities and function, scored on a 0-52 point scale, with greater scores indicating a better fatigue-related quality of life. The change from baseline in FACIT-Fatigue score will be presented.
Percentage of Diagnostic Assay Positive (Dx+) Participants Achieving Clinical Remission Per MMS at Week 12 | Week 12
  Dx+ participants are those who meet protocol-specific diagnostic assay criteria during screening. The MMS is a composite score of UC disease activity on a scale of increasing severity from 0-9, calculated by summing three subscores: ES, scored on a scale of increasing severity from 0 (normal or inactive disease) to 3 (severe disease, such as spontaneous bleeding or ulceration); SFS, scored on a scale of increasing frequency from 0 (normal number of stools) to 3 (≥5 stools more than normal per day for the participant); and RBS, scored on a scale of increasing severity from 0 (no blood seen) to 3 (blood alone passed). Clinical Remission is defined as an ES of 0 or 1, RBS of 0, and SFS of 0 or 1 and not greater than the baseline SFS.
Percentage of Dx+ Participants With Endoscopic Improvement at Week 12 | Week 12
  Dx+ participants are those who meet protocol-specific diagnostic assay criteria during screening. Endoscopic improvement is defined as ES of 0 or 1. The ES measures UC severity based on endoscopy on a 0-3 scale of increasing severity.
Study 1: Percentage of Participants Achieving Histologic-Endoscopic Remission (HER) at Week 12 | Week 12
  HER is defined as a Geboes score of less than 2 and ES of 0 or 1. The Geboes score is a histologic grading system for inflammation in UC with scores ranging from 0 to 5.4, with higher scores indicating more severe inflammation. ES measures UC severity based on endoscopy, scored from 0 (normal or inactive disease) to 3 (severe disease, such as spontaneous bleeding or ulceration).
Study 1: Percentage of Participants with Endoscopic Improvement at Week 52 | Week 52
  Endoscopic improvement is defined as ES of 0 or 1. The ES measures UC severity based on endoscopy on a 0-3 scale of increasing severity.
Study 1: Percentage of Participants Achieving Corticosteroid-Free Clinical Remission Per MMS at Week 52 | Week 52
  The Modified Mayo Score (MMS) is a composite score of ulcerative colitis (UC) disease activity on a scale of increasing severity from 0-9, calculated by summing three subscores: Endoscopic subscore (ES), scored on a scale of increasing severity from 0 (normal or inactive disease) to 3 (severe disease, such as spontaneous bleeding or ulceration); Stool frequency subscore (SFS), scored on a scale of increasing frequency from 0 (normal number of stools) to 3 (≥5 stools more than normal per day for the participant); and rectal bleeding subscore (RBS), scored on a scale of increasing severity from 0 (no blood seen) to 3 (blood alone passed). Corticosteroid-free clinical remission is defined as an ES of 0 or 1, RBS of 0, and SFS of 0 or 1 and not greater than the baseline SFS, and no corticosteroid use for ≥90 days before Week 52.
Study 1: Percentage of Participants Achieving HEMI at Week 52 | Week 52
  HEMI is defined as a Geboes score of 3.1 or less and ES of 0 or 1. The Geboes score is a histologic grading system for inflammation in UC with scores ranging from 0 to 5.4, with higher scores indicating more severe inflammation. ES measures UC severity based on endoscopy, scored from 0 (normal or inactive disease) to 3 (severe disease, such as spontaneous bleeding or ulceration).
Study 1: Percentage of Participants Achieving Clinical Remission Per pMMS at Week 52 | Week 52
  pMMS is a composite score of UC disease activity on a scale of increasing severity from 0-6, calculated by summing two subscores: SFS, scored from 0 (normal number of stools) to 3 (≥5 stools more than normal per day for the participant); RBS, scored from 0 (no blood seen) to 3 (blood alone passed). Clinical remission per pMMS is defined as an RBS of 0 and SFS of ≤1.
Study 1: Percentage of Participants Achieving Sustained Clinical Remission Per MMS at Both Week 12 and Week 52 | Week 12 and Week 52
  The MMS is a composite score of UC disease activity on a scale of increasing severity from 0-9, calculated by summing three subscores: ES, scored on a scale of increasing severity from 0 (normal or inactive disease) to 3 (severe disease, such as spontaneous bleeding or ulceration); SFS, scored on a scale of increasing frequency from 0 (normal number of stools) to 3 (≥5 stools more than normal per day for the participant); and RBS, scored on a scale of increasing severity from 0 (no blood seen) to 3 (blood alone passed). Sustained clinical remission is defined as an ES of 0 or 1, RBS of 0, and SFS of 0 or 1 and not greater than the baseline SFS, at both Week 12 and Week 52.
Study 1: Percentage of Participants Reporting No Bowel Urgency at Week 52 | Week 52
  Bowel urgency is measured using an NRS, which rates bowel urgency on a 0-11 scale of increasing severity. Resolution is defined as a score of 0 or 1 in participants who had a baseline score of 3 or more.
Study 1: Percentage of Participants Reporting No Abdominal Pain at Week 52 | Week 52
  Abdominal pain is measured on a 0-4 NRS of increasing pain severity. Absence of abdominal pain is defined as a rating of 0.
Study 1: Percentage of Participants With Endoscopic Remission at Week 52 | Week 52
  ES measures UC severity based on endoscopy, scored from 0 (normal or inactive disease) to 3 (severe disease, such as spontaneous bleeding or ulceration). Endoscopic remission is defined as an ES of 0.
Study 1: Percentage of Participants with Sustained Endoscopic Improvement at Both Week 12 and Week 52 | Week 12 and Week 52
  Sustained endoscopic improvement is defined as an ES of 0 or 1 at both Week 12 and Week 52. The ES measures UC severity based on endoscopy on a 0-3 scale of increasing severity.
Study 1: Percentage of Participants Achieving HER at Week 52 | Week 52
  HER is defined as a Geboes score of less than 2 and ES of 0 or 1. The Geboes score is a histologic grading system for inflammation in UC with scores ranging from 0 to 5.4, with higher scores indicating more severe inflammation. ES measures UC severity based on endoscopy, scored from 0 (normal or inactive disease) to 3 (severe disease, such as spontaneous bleeding or ulceration).
Study 1: Percentage of Participants Achieving IBDQ Remission at Week 52 | Week 52
  The IBDQ measures health related quality of life in subjects with inflammatory bowel disease. It consists of 32 questions each with a graded response of 1 (worst) to 7 (best). The score ranges from 32 to 224. IBDQ remission is defined as a score of at least 170.
Study 1: Change from Baseline in FACIT-Fatigue Score at Week 52 | Baseline and Week 52
  The FACIT-Fatigue is a 13-item measure that assesses self-reported fatigue and its impact upon daily activities and function, scored on a 0-52 point scale, with greater scores indicating a better fatigue-related quality of life. The change from baseline in FACIT-Fatigue score will be presented.
Study 1: Percentage of Dx+ Participants Achieving Clinical Remission Per MMS at Week 52 | Week 52
  Dx+ participants are those who meet protocol-specific diagnostic assay criteria during screening. The MMS is a composite score of UC disease activity on a scale of increasing severity from 0-9, calculated by summing three subscores: ES, scored on a scale of increasing severity from 0 (normal or inactive disease) to 3 (severe disease, such as spontaneous bleeding or ulceration); SFS, scored on a scale of increasing frequency from 0 (normal number of stools) to 3 (≥5 stools more than normal per day for the participant); and RBS, scored on a scale of increasing severity from 0 (no blood seen) to 3 (blood alone passed). Clinical Remission is defined as an ES of 0 or 1, RBS of 0, and SFS of 0 or 1 and not greater than the baseline SFS.
Study 1: Percentage of Dx+ Participants With Endoscopic Improvement at Week 52 | Week 52
  Dx+ participants are those who meet protocol-specific diagnostic assay criteria during screening. Endoscopic improvement is defined as ES of 0 or 1. The ES measures UC severity based on endoscopy on a 0-3 scale of increasing severity.
Study 2: Percentage of Participants With One or More AEs | Up to approximately 12 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who experience an AE will be reported.
Study 2: Percentage of Participants Who Discontinued Study Intervention Due to an AE | Up to approximately 12 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinue study treatment due to an AE will be reported.
Study 2: Percentage of Participants with Clinical Response Per pMMS at Week 2 | Week 2
  pMMS is a composite score of UC disease activity on a scale of increasing severity from 0-6, calculated by summing two subscores: SFS, scored from 0 (normal number of stools) to 3 (≥5 stools more than normal per day for the participant); RBS, scored from 0 (no blood seen) to 3 (blood alone passed). Clinical response is defined as pMMS reduction of 1 or more points and 30% or more, plus a reduction of 1 or more points in RBS or an absolute RBS of 0 or 1.
Study 2: Percentage of Participants With Endoscopic Improvement at Week 12 | Week 12
  Endoscopic improvement is defined as Mayo endoscopic subscore (ES) of 0 or 1. The ES measures UC severity based on endoscopy on a 0-3 scale of increasing severity.
Study 2: Percentage of Participants Achieving a Clinical Response Per MMS at Week 12 | Week 12
  The MMS is a composite score of UC disease activity on a scale of increasing severity from 0-9, calculated by summing three subscores: ES, scored on a scale of increasing severity from 0 (normal or inactive disease) to 3 (severe disease, such as spontaneous bleeding or ulceration); SFS, scored on a scale of increasing frequency from 0 (normal number of stools) to 3 (≥5 stools more than normal per day for the participant); and RBS, scored on a scale of increasing severity from 0 (no blood seen) to 3 (blood alone passed). Clinical response is defined as an MMS reduction of 2 or more points and 30% or more, plus a reduction of more than 1 point in RBS or an absolute RBS of 0 or 1.
Study 2: Percentage of Participants Achieving HEMI at Week 12 | Week 12
  HEMI is defined as a Geboes score of 3.1 or less and ES of 0 or 1. The Geboes score is a histologic grading system for inflammation in UC with scores ranging from 0 to 5.4, with higher scores indicating more severe inflammation. ES measures UC severity based on endoscopy, scored from 0 (normal or inactive disease) to 3 (severe disease, such as spontaneous bleeding or ulceration).
Study 2: Percentage of Participants Achieving Clinical Remission Per pMMS at Week 12 | Week 12
  pMMS is a composite score of UC disease activity on a scale of increasing severity from 0-6, calculated by summing two subscores: SFS, scored from 0 (normal number of stools) to 3 (≥5 stools more than normal per day for the participant); RBS, scored from 0 (no blood seen) to 3 (blood alone passed). Clinical remission per pMMS is defined as an RBS of 0 and SFS of ≤1.
Study 2: Percentage of Participants With Endoscopic Remission at Week 12 | Week 12
  ES measures UC severity based on endoscopy, scored from 0 (normal or inactive disease) to 3 (severe disease, such as spontaneous bleeding or ulceration). Endoscopic remission is defined as an ES of 0.
Study 2: Percentage of Participants Reporting No Bowel Urgency at Week 12 | Week 12
  Bowel urgency is measured using a numeric rating scale (NRS), which rates bowel urgency on a 0-11 scale of increasing severity.
Study 2: Percentage of Participants Reporting No Abdominal Pain at Week 12 | Week 12
  Abdominal pain is measured on a 0-4 NRS of increasing pain severity. Absence of abdominal pain is defined as a rating of 0.
Study 2: Percentage of Participants Achieving IBDQ Remission at Week 12 | Week 12
  The IBDQ measures health related quality of life in subjects with inflammatory bowel disease. It consists of 32 questions each with a graded response of 1 (worst) to 7 (best). The score ranges from 32 to 224. IBDQ remission is defined as a score of at least 170.
Study 2: Change from Baseline in FACIT-Fatigue Score at Week 12 | Baseline and Week 12
  The FACIT-Fatigue is a 13-item measure that assesses self-reported fatigue and its impact upon daily activities and function, scored on a 0-52 point scale, with greater scores indicating a better fatigue-related quality of life. The change from baseline in FACIT-Fatigue score will be presented.
Study 2: Percentage of Participants Achieving HER at Week 12 | Week 12
  HER is defined as a Geboes score of less than 2 and ES of 0 or 1. The Geboes score is a histologic grading system for inflammation in UC with scores ranging from 0 to 5.4, with higher scores indicating more severe inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (476):
- United States (76):
  - Digestive Health Specialists ( Site 0135), Dothan, Alabama
  - IMC-Gulf Coast Gastroenterology ( Site 0157), Fairhope, Alabama
  - Research Solutions of Arizona ( Site 3816), Litchfield Park, Arizona
  - One of a Kind Clinical Research Center ( Site 3852), Scottsdale, Arizona
  - GI Alliance - Sun City ( Site 0103), Sun City, Arizona
  - Clinnova Research ( Site 3803), Anaheim, California
  - Southern California Research Center ( Site 3828), Coronado, California
  - UCSD - Altman Clinical and Translational Research Institute (ACTRI) ( Site 0113), La Jolla, California
  - Cedars-Sinai Medical Center ( Site 0119), Los Angeles, California
  - University of California, Irvine (UCI) Health - UC Irvine Medical Center ( Site 3851), Orange, California
  - University of Colorado Anschutz Medical Campus-Division of Gastroenterology and Hepatology ( Site 0172), Aurora, Colorado
  - Peak Gastroenterology Associates ( Site 0116), Colorado Springs, Colorado
  - South Denver Gastroenterology, PC ( Site 3849), Englewood, Colorado
  - Rocky Mountain Gastroenterology/Topography Health ( Site 3838), Littleton, Colorado
  - Connecticut Clinical Research Institute ( Site 0126), Bristol, Connecticut
  - Medical Research Center of Connecticut ( Site 0151), Hamden, Connecticut
  - Yale University School of Medicine-Digestive Disease ( Site 0163), New Haven, Connecticut
  - Emerson Clinical Research Institute ( Site 3820), Washington D.C., District of Columbia
  - Gastroenterology Consultants of Clearwater ( Site 0152), Clearwater, Florida
  - University of Florida College of Medicine-Gastroenterology ( Site 3821), Gainesville, Florida
  - Nature Coast Clinical Research - Inverness ( Site 3806), Inverness, Florida
  - Central Florida Gastro Research ( Site 0124), Kissimmee, Florida
  - Research Associates of South Florida - Miami - Southwest 8th Street ( Site 3810), Miami, Florida
  - Orlando Health ( Site 0145), Orlando, Florida
  - USF Health ( Site 0169), Tampa, Florida
  - Emory University School of Medicine ( Site 3818), Atlanta, Georgia
  - Atlanta Gastroenterology Associates - Peachtree Dunwoody ( Site 0115), Atlanta, Georgia
  - Atlanta Center for Gastroenterology ( Site 0155), Decatur, Georgia
  - University of Chicago Medical Center ( Site 0134), Chicago, Illinois
  - GI Alliance - Glenview ( Site 0168), Glenview, Illinois
  - GI ALLIANCE - GURNEE ( Site 0107), Gurnee, Illinois
  - Iowa Digestive Disease Center ( Site 0123), Clive, Iowa
  - University of Louisville Hospital-Clinical Trials Unit ( Site 0165), Louisville, Kentucky
  - Baton Rouge General Medical Center - Bluebonnet ( Site 0112), Baton Rouge, Louisiana
  - Tulane University School of Medicine-Gastroenterology and Hepatology ( Site 0154), New Orleans, Louisiana
  - Walter Reed National Military Medical Center ( Site 0121), Bethesda, Maryland
  - Woodholme Gastroenterology Associates-Woodholme Gastroenterology Associates ( Site 3835), Glen Burnie, Maryland
  - Massachusetts General Hospital-Crohn's and Colitis Center ( Site 0132), Boston, Massachusetts
  - University of Michigan ( Site 0143), Ann Arbor, Michigan
  - Clinical Research Institute of Michigan, LLC ( Site 0108), Clinton Township, Michigan
  - Michigan Center of Medical Research (MICHMER) ( Site 3850), Farmington Hills, Michigan
  - Clinical Research Institute of Michigan, LLC ( Site 0150), Troy, Michigan
  - Huron Gastroenterology ( Site 3836), Ypsilanti, Michigan
  - Mayo Clinic in Rochester, Minnesota ( Site 0147), Rochester, Minnesota
  - BVL Research - Kansas ( Site 3847), Liberty, Missouri
  - Washington University School of Medicine ( Site 0129), St Louis, Missouri
  - Circuit Clinical /Middletown Medical PC ( Site 3831), Middletown, New York
  - NYU Langone Health - Inflammatory Bowel Disease Center (IBD) ( Site 3846), New York, New York
  - Lenox Hill Hospital ( Site 0128), New York, New York
  - New York Gastroenterology Associates ( Site 0159), New York, New York
  - University of North Carolina Medical Center ( Site 0140), Chapel Hill, North Carolina
  - Carolina Digestive Diseases and Endoscopy Center ( Site 3809), Greenville, North Carolina
  - Hospital of the University of Pennsylvania ( Site 0170), Philadelphia, Pennsylvania
  - University Gastroenterology ( Site 0164), Providence, Rhode Island
  - Gastroenterology Associates of Orangeburg ( Site 0149), Orangeburg, South Carolina
  - Vanderbilt Inflammatory Bowel Disease Clinic ( Site 0131), Nashville, Tennessee
  - Quality Medical Research ( Site 3807), Nashville, Tennessee
  - GI Alliance - Garland ( Site 0109), Garland, Texas
  - Baylor College of Medicine Medical Center ( Site 3812), Houston, Texas
  - The University of Texas Health Science Center at Houston-Internal Medicine-Division of Gastroentero ( Site 0144), Houston, Texas
  - Clinical Trial Network ( Site 3819), Houston, Texas
  - GI Alliance - Lubbock ( Site 0167), Lubbock, Texas
  - Caprock Gastro Research ( Site 0101), Lubbock, Texas
  - GI Alliance: Mansfield ( Site 0161), Mansfield, Texas
  - CARTA - Clinical Associates In Research Therapeutics Of America ( Site 0122), San Antonio, Texas
  - Southern Star Research Institute ( Site 0106), San Antonio, Texas
  - GI Alliance - San Marcos ( Site 0130), San Marcos, Texas
  - GI Alliance - Southlake ( Site 0104), Southlake, Texas
  - Tyler Research Institute ( Site 0105), Tyler, Texas
  - Texas Digestive Disease Consultants ( Site 0136), Webster, Texas
  - Velocity Clinical Research, Salt Lake City ( Site 3801), West Jordan, Utah
  - Richmond VA Medical Center ( Site 3845), Richmond, Virginia
  - Washington Gastroenterology - Bellevue ( Site 3844), Bellevue, Washington
  - University of Washington Medical Center - Montlake ( Site 0137), Seattle, Washington
  - Washington Gastroenterology - Tacoma ( Site 0102), Tacoma, Washington
  - MEDICAL COLLEGE OF WISCONSIN ( Site 0141), Milwaukee, Wisconsin
- Argentina (4):
  - Centro de Investigaciones Médicas Mar del Plata ( Site 2101), Mar del Plata, Buenos Aires
  - CER medical Institute-Gastroenterology ( Site 2110), Quilmes, Buenos Aires F.D.
  - Hospital Provincial del Centenario ( Site 2108), Rosario, Santa Fe Province
  - C.I.C.E. 9 de Julio-CICE 9 DE JULIO ( Site 2103), San Miguel de Tucumán, Tucumán Province
- Australia (8):
  - Nepean Hospital-Gastroenterology/Hepatology ( Site 2501), Kingswood, New South Wales
  - Concord Repatriation General Hospital-Gastroenterology and Liver Services ( Site 2508), Sydney, New South Wales
  - Royal Brisbane and Women's Hospital ( Site 2500), Brisbane, Queensland
  - Mater Misericordiae Limited-Gastroenterology ( Site 2506), Brisbane, Queensland
  - Royal Adelaide Hospital-Gastroenterology/Hepatology ( Site 2504), Adelaide, South Australia
  - Monash Health-Gastroenterology ( Site 2505), Clayton, Victoria
  - The Alfred Hospital-Gastroenterology ( Site 2503), Melbourne, Victoria
  - St Vincent's Hospital ( Site 2510), Melbourne, Victoria
- Austria (3):
  - Universitaetsklinik fuer Innere Medizin I Innsbruck ( Site 0200), Innsbruck, Tyrol
  - Medizinische Universität Wien-Klinik für Innere Medizin III - Abteilung für Gastroenterologie und H ( Site 0202), Vienna, Vienna
  - Uniklinikum Salzburg-Innere Medizin I ( Site 0201), Salzburg
- Belgium (2):
  - UZ Gent ( Site 0300), Ghent, Oost-Vlaanderen
  - UZ Leuven-Gastroenterology - Inflammatory Bowel Disease ( Site 0301), Leuven, Vlaams-Brabant
- Brazil (6):
  - L2IP - Instituto de Pesquisas Clínicas ( Site 5104), Brasília, Federal District
  - Endogastro Clínica de Gastroenterologia e Endoscopia Digestiva Lida - Galileo Pesquisa Clínica ( Site 5100), Juiz de Fora, Minas Gerais
  - Hospital Moinhos de Vento ( Site 5108), Porto Alegre, Rio Grande do Sul
  - Pesquisare Saude ( Site 5112), Santo André, São Paulo
  - Centro de Pesquisa Kaiser - CEPEK ( Site 5103), São José do Rio Preto, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto ( Site 5107), São José do Rio Preto, São Paulo
- Bulgaria (9):
  - MC Velingrad 2017 EOOD ( Site 0406), Velingrad, Pazardzhik
  - "Diagnostic - Consultative Center XX - Sofia" EOOD ( Site 0407), Sofia, Sofia (stolitsa)
  - Medconsult Pleven ( Site 0410), Pleven
  - DKC V - Plovdiv ( Site 0402), Plovdiv
  - MC Rusemed ( Site 0408), Rousse
  - MHAT Hadzhi Dimitar-Gastroenterology ( Site 0403), Sliven
  - Diagnostic Consultative Center 22 - Sofia ( Site 0401), Sofia
  - 4th MHAT ( Site 0409), Sofia
  - Medica Plus Medical Center ( Site 0404), Veliko Tarnovo
- Canada (17):
  - Heritage Medical Research Clinic ( Site 0004), Calgary, Alberta
  - Gastroenterology and internal medicine research institute ( Site 0010), Edmonton, Alberta
  - Prairie Institute of Liver and Luminal Advanced Research ( Site 0013), Lethbridge, Alberta
  - Fraser Clinical Trials Inc. ( Site 0019), New Westminster, British Columbia
  - G.I.R.I. GI Research Institute Foundation ( Site 0001), Vancouver, British Columbia
  - Private Practice - Dr. Bruce Musgrave ( Site 0011), Kentville, Nova Scotia
  - Barrie GI Associates ( Site 0012), Barrie, Ontario
  - University Hospital - London Health Sciences Centre ( Site 0002), London, Ontario
  - London Health Sciences Centre ( Site 0007), London, Ontario
  - West GTA Research Inc. ( Site 0017), Mississauga, Ontario
  - ABP Research Services Corp. ( Site 0016), Ontario, Ontario
  - Toronto Immune & Digestive Health Institute ( Site 0005), Toronto, Ontario
  - Toronto Digestive Disease Associates ( Site 0006), Vaughan, Ontario
  - Centre Intégré de Santé et Service Sociaux de Chaudière-Appalaches ( Site 0015), Lévis, Quebec
  - Centre Hospitalier de l Universite de Montreal - CHUM ( Site 0018), Montreal, Quebec
  - Montreal General Hospital ( Site 0003), Montreal, Quebec
  - Diex Recherche Quebec ( Site 0008), Québec, Quebec
- Chile (8):
  - Clinical Research Chile SpA ( Site 2201), Valdivia, Los Ríos Region
  - Centro de Estudios Clínicos SAGA-CECSAGA ( Site 2203), Santiago, Region M. de Santiago
  - FALP-UIDO ( Site 2208), Santiago, Region M. de Santiago
  - Clínica Universidad de Los Andes ( Site 2202), Santiago, Region M. de Santiago
  - Clínica Alemana de Santiago ( Site 2209), Santiago, Region M. de Santiago
  - Clínica MEDS La Dehesa ( Site 2207), Santiago, Region M. de Santiago
  - CECIM ( Site 2200), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile-CICUC ( Site 2205), Santiago, Region M. de Santiago
- China (38):
  - The First Affiliated Hospital of Anhui Medical University ( Site 3957), Hefei, Anhui
  - Anhui Provincial Hospital ( Site 3947), Hefei, Anhui
  - Beijing Friendship Hospital Affiliate of Capital University ( Site 3923), Beijing, Beijing Municipality
  - Peking University Third Hospital ( Site 3909), Beijing, Beijing Municipality
  - Beijing Luhe Hospital Capital Medical University ( Site 3911), Beijing, Beijing Municipality
  - Chongqing University Three Gorges Hospital ( Site 3928), Chongqing, Chongqing Municipality
  - The First Affiliated Hospital Of Fujian Medical University ( Site 3904), Fuzhou, Fujian
  - The First Affiliated hospital of Xiamen University-Gastroenterology ( Site 3954), Xiamen, Fujian
  - Dongguan People's Hospital-Gastroenterology department ( Site 3944), Dongguan, Guangdong
  - Guangzhou Medical University 2nd Hospital ( Site 3908), Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital-Gastroenterology ( Site 3914), Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University ( Site 3906), Guangzhou, Guangdong
  - Huizhou Municipal Central Hospital ( Site 3917), Huizhou, Guangdong
  - Yuebei People's Hospital Guangdong ( Site 3948), Shaoguan, Guangdong
  - The University of Hong Kong-Shenzhen Hospital ( Site 3955), Shenzhen, Guangdong
  - Shenzhen Hospital of Southern Medical University ( Site 3905), Shenzhen, Guangdong
  - The Second Hospital of Hebei Medical University ( Site 3934), Shijiazhuang, Hebei
  - The Second Affiliated Hospital of Zhengzhou University ( Site 3935), Zhengzhou, Henan
  - Taihe Hospital ( Site 3941), Shiyan, Hubei
  - The Central Hospital of Wuhan ( Site 3939), Wuhan, Hubei
  - Renmin Hospital of Wuhan University ( Site 3912), Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University ( Site 3930), Changsha, Hunan
  - Changzhou No.2 People's Hospital ( Site 3950), Changzhou, Jiangsu
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School ( Site 3900), Nanjing, Jiangsu
  - Zhongda Hospital Southeast University ( Site 3919), Nanjing, Jiangsu
  - Wuxi People's Hospital ( Site 3920), Wuxi, Jiangsu
  - The First Affiliated Hospital of Nanchang University ( Site 3926), Nanchang, Jiangxi
  - Tangdu Hospital of Fourth Military Medical University of Chinese People's Liberation Army ( Site 3929), Xi'an, Shaanxi
  - Binzhou Medical University Hospital ( Site 3953), Binzhou, Shandong
  - Taian City Central Hospital-gastroenterology department ( Site 3946), Taian, Shandong
  - Ruijin Hospital Shanghai Jiaotong University School of Medicine-Gastroneterology ( Site 3903), Shanghai, Shanghai Municipality
  - Shanghai East Hospital ( Site 3922), Shanghai, Shanghai Municipality
  - Renji Hospital Shanghai Jiao Tong University School of Medicine ( Site 3915), Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University ( Site 3951), Chengdu, Sichuan
  - Tianjin Medical University General Hospital ( Site 3945), Tianjin, Tianjin Municipality
  - The First Teaching Hospital of Xinjiang Medical University. ( Site 3937), Ürümqi, Xinjiang
  - First Affiliated Hospital of Kunming Medical University ( Site 3925), Kunming, Yunnan
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine-GI Medicine ( Site 3916), Hangzhou, Zhejiang
- Colombia (7):
  - Clínica las Américas ( Site 2318), Medellín, Antioquia
  - Clinica Medellin S.A ( Site 2317), Medellín, Antioquia
  - Clinica Somer-Unidad de Investigacion y Docencia ( Site 2303), Rionegro, Antioquia
  - Clinica de la Costa S.A.S. ( Site 2305), Barranquilla, Atlántico
  - Fundacion Santa Fe de Bogota ( Site 2316), Bogota, Cundinamarca
  - Oncologos del Occidente ( Site 2310), Pereira, Risaralda Department
  - Fundación Valle del Lili ( Site 2307), Cali, Valle del Cauca Department
- Croatia (6):
  - Klinička bolnica Merkur ( Site 0505), Zagreb, City of Zagreb
  - Klinički bolnički centar Zagreb ( Site 0501), Zagreb, City of Zagreb
  - Poliklinika Bates ( Site 0504), Zagreb, City of Zagreb
  - Poliklinika Solmed ( Site 0502), Zagreb, City of Zagreb
  - Poliklinika Borzan ( Site 0500), Osijek, County of Osijek-Baranja
  - Klinički Bolnički Centar Split ( Site 0503), Split, Split-Dalmatia County
- Czechia (4):
  - Vojenská Nemocnice Brno-Internal department ( Site 0605), Brno, Brno-mesto
  - Nemocnice Slany ( Site 0601), Slaný, Central Bohemia
  - Institut Klinicke a Experimentalni Mediciny-Klinika hepatogastroentrologie ( Site 0604), Prague, Praha 4
  - Hepato-Gastroenterologie HK ( Site 0602), Hradec Králové
- CEMDOE - Centro Médico de Diabetes, Obesidad y Especialidades ( Site 3601), Santo Domingo, Nacional, Dominican Republic
- Finland (3):
  - Tampereen yliopistollinen sairaala ( Site 4300), Tampere, Pirkanmaa
  - Pohjois-Karjalan keskussairaala ( Site 4302), Joensuu, Pohjois-Karjala
  - Turku University Hospital ( Site 4301), Turku, Southwest Finland
- France (18):
  - Centre Hospitalier Universitaire de Nice - Hôpital l'Archet ( Site 0706), Nice, Alpes-Maritimes
  - CHU Bordeaux Haut-Leveque-Service d'Hépato-gastroentérologie ( Site 0700), Pessac, Aquitaine
  - Assistance Publique Hôpitaux de Marseille - Hôpital Nord ( Site 0714), Marseille, Bouches-du-Rhone
  - Centre Hospitalier Universitaire de Reims - Hôpital Robert Debré ( Site 0705), Reims, Champagne-Ardenne
  - CHU Besançon ( Site 0710), Besançon, Doubs
  - C.H.U. de Nimes. Hopital Caremeau ( Site 0718), Nîmes, Gard
  - Hopital Beaujon ( Site 0716), Clichy, Hauts-de-Seine
  - CMC Ambroise Paré Hartmann - Institut des MICI ( Site 0709), Neuilly-sur-Seine, Hauts-de-Seine
  - Clinique des Cèdres ( Site 0719), Échirolles, Isere
  - CHU SAINT ELOI ( Site 0711), Montpellier, Languedoc-Roussillon
  - Centre Hospitalier Régional Universitaire de Nancy - Hôpitaux de Brabois ( Site 0708), Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Centre Hospitalier Universitaire de Nantes - L' Hopital l'hôtel-Dieu ( Site 0701), Nantes, Pays de la Loire Region
  - centre hospitalier lyon sud ( Site 0707), Pierre-Bénite, Rhone
  - CHU d'Amiens-Picardie - Hôpital Sud-Hepato-gastroentérology ( Site 0712), Amiens, Somme
  - Hopital Henri Mondor ( Site 0717), Créteil, Val-de-Marne
  - Hôpitaux Universitaires Paris Sud - Hôpital Bicêtre ( Site 0715), Le Kremlin-Bicêtre, Val-de-Marne
  - Hôpital Saint Antoine ( Site 0703), Paris
  - Hôpital Saint-Louis ( Site 0702), Paris
- Georgia (4):
  - LTD High Technology Hospital Medcenter ( Site 0802), Batumi, Adjara
  - Caucasus Medical Centre ( Site 0801), Tbilisi, Adjara
  - Caraps Medline ( Site 0803), Tbilisi
  - New Hospitals ( Site 0800), Tbilisi
- Germany (14):
  - Universitaetsklinikum Ulm. ( Site 0902), Ulm, Baden-Wurttemberg
  - MVZ Dachau ( Site 0918), Dachau, Bavaria
  - Klinikum der Universität München Großhadern-Medizinische Klinik und Poliklinik II ( Site 0907), Munich, Bavaria
  - Agaplesion Markus Krankenhaus ( Site 0904), Frankfurt am Main, Hesse
  - Medizinische Hochschule Hannover ( Site 0913), Hanover, Lower Saxony
  - Klinikum Lüneburg ( Site 0908), Lüneburg, Lower Saxony
  - Stadtische Kliniken Duisburg, Abtlg. Innere Medizin ( Site 0916), Duisburg, North Rhine-Westphalia
  - Gastroenterologische Gemeinschaftspraxis Minden ( Site 0911), Minden, North Rhine-Westphalia
  - Medizinisches Versorgungszentrum Portal 10 ( Site 0914), Münster, North Rhine-Westphalia
  - St. Marien und St. Annastift Krankenhaus ( Site 0901), Ludwighafen Am Rhein, Rhineland-Palatinate
  - Universitätsklinikum Leipzig ( Site 0909), Leipzig, Saxony
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel ( Site 0903), Kiel, Schleswig-Holstein
  - Charité Campus Virchow-Klinikum ( Site 0906), Berlin
  - Universitätsklinikum Brandenburg an der Havel ( Site 0905), Brandenburg
- Greece (5):
  - Evangelismos General Hospital of Athens ( Site 4001), Athens, Attica
  - THORACIC GENERAL HOSPITAL OF ATHENS "I SOTIRIA"-3rd Dept of Internal Medicine and Laboratory, Oncol ( Site 4000), Athens, Attica
  - General Hospital of Nikaia-Piraeus "Agios Panteleimon" ( Site 4006), Nikaia Piraeus, Attica
  - Ippokrateio General Hospital of Thessaloniki ( Site 4004), Thessaloniki, Central Macedonia
  - University General Hospital of Heraklion-GASTROENTEROLOGY & HEPATOLOGY ( Site 4003), Heraklion, Crete
- Hungary (10):
  - Mohácsi Kórház ( Site 1008), Mohács, Baranya
  - Békés Megyei Központi Kórház Dr. Réthy Pál Tagkórház-4. Belgyogyaszat Gasztroenterologia ( Site 1007), Békéscsaba, Bekescsaba
  - Csőszi Endoszkópos KFT ( Site 1001), Kecskemét, Bács-Kiskun county
  - Heves Vármegyei Markhot Ferenc Oktatókórház és Rendelőintézet ( Site 1012), Eger, Heves County
  - Gyöngyösi Bugát Pál Kórház ( Site 1011), Gyöngyös, Heves County
  - Komarom-Esztergom Varmegyei Szent Borbala Korhaz ( Site 1010), Tatabánya, Komárom-Esztergom
  - VeszLife Magánklinika ( Site 1002), Veszprém, Veszprém megye
  - Synexus Magyarorszag Kft. (Budapest DRS) ( Site 1009), Budapest
  - Semmelweis Egyetem ( Site 1006), Budapest
  - Pannónia Magánorvosi Centrum ( Site 1004), Budapest
- Israel (9):
  - Emek Medical Center ( Site 1106), Afula
  - Barzilai Medical Center ( Site 1109), Ashkelon
  - Rambam Health Care Campus ( Site 1101), Haifa
  - Bnai Zion Medical Center ( Site 1103), Haifa
  - Edith Wolfson Medical Center ( Site 1104), Holon
  - Shaare Zedek Medical Center ( Site 1108), Jerusalem
  - Meir Medical Center. ( Site 1102), Kfar Saba
  - Rabin Medical Center ( Site 1107), Petah Tikva
  - Sheba Medical Center ( Site 1100), Ramat Gan
- Italy (16):
  - Policlinico Universitario Monserrato-SC Gastroenterologia ( Site 1207), Monserrato, Cagliari
  - IRCCS Casa Sollievo della Sofferenza ( Site 1213), San Giovanni Rotondo, Foggia
  - Fondazione Policlinico Tor Vergata ( Site 1209), Rome, Lazio
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico-Gastroenterology and Endoscopy Unit ( Site 1202), Milan, Lombardy
  - Istituto Clinico Humanitas-IBD center ( Site 1201), Rozzano, Lombardy
  - Ospedale Di Circolo-U.O.C. di Gastroenterologia ed Endoscopia Digestiva ( Site 1216), Rho, Milano
  - A.O.R.N. Ospedale dei Colli - Monaldi V. ( Site 1217), Naples, Napoli
  - Azienda Ospedaliera San Camillo Forlanini ( Site 1204), Rome, Roma
  - Fatebenefratelli Isola Tiberina - Gemelli Isola ( Site 1214), Rome, Roma
  - Az. Osp. Ospedali Riuniti VILLA SOFIA-CERVELLO-U.O.S.D. Malattie Infiammatorie Croniche Intestinali ( Site 1210), Palermo, Sicily
  - Azienda Ospedale - Università Padova-Surgery Oncology and Gastroenterology ( Site 1211), Padua, Veneto
  - Ospedale Sacro Cuore Don G. Calabria ( Site 1212), Negrar, Verona
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola ( Site 1208), Bologna
  - ASST Fatebenefratelli Sacco-UOC Gastroenterologia ( Site 1200), Milan
  - Ospedale San Raffaele-Gastroenterology and Gastrointestinal Endoscopy ( Site 1205), Milan
  - Fondazione IRCCS Policlinico San Matteo-General Medicine ( Site 1206), Pavia
- Japan (54):
  - Aichi Medical University Hospital ( Site 2841), Nagakute, Aichi-ken
  - Tokatsu Tsujinaka Hospital ( Site 2832), Abiko, Chiba
  - Tsujinaka Hospital - Kashiwanoha ( Site 2802), Kashiwa, Chiba
  - Toho University Sakura Medical Center ( Site 2805), Sakura, Chiba
  - Ehime Prefectural Central Hospital ( Site 2868), Matsuyama, Ehime
  - Kitakyushu Municipal Medical Center ( Site 2873), Kitakyushu, Fukuoka
  - Kurume University Hospital ( Site 2846), Kurume, Fukuoka
  - Gunma University Hospital ( Site 2850), Maebashi, Gunma
  - National Hospital Organization Fukuyama Medical Center ( Site 2831), Fukuyama, Hiroshima
  - Asahikawa City Hospital ( Site 2840), Asahikawa, Hokkaido
  - Asahikawa Medical University Hospital ( Site 2815), Asahikawa, Hokkaido
  - Sapporo Tokushukai Hospital ( Site 2808), Sapporo, Hokkaido
  - Sapporo Medical University Hospital ( Site 2829), Sapporo, Hokkaido
  - Medical Corporation Sapporo IBD Clinic ( Site 2842), Sapporo, Hokkaido
  - Sapporohigashi Tokushukai Hospital ( Site 2860), Sapporo, Hokkaido
  - Hyogo Medical University Hospital ( Site 2830), Nishinomiya, Hyōgo
  - Hitachi General Hospital ( Site 2856), Hitachi, Ibaraki
  - Ishikawa Prefectural Central Hospital ( Site 2835), Kanazawa, Ishikawa-ken
  - Kanazawa University Hospital ( Site 2839), Kanazawa, Ishikawa-ken
  - Iwate Medical University Uchimaru Medical Center ( Site 2833), Morioka, Iwate
  - Gokeikai Ofuna Chuo Hospital ( Site 2801), Kamakura, Kanagawa
  - St. Marianna University Hospital ( Site 2852), Kawasaki, Kanagawa
  - Matsushima Hospital ( Site 2822), Yokohama, Kanagawa
  - Yokohama City University Medical Center ( Site 2865), Yokohama, Kanagawa
  - Mie University Hospital ( Site 2838), Tsu, Mie-ken
  - Sai Gastroenterology/Proctology Clinic ( Site 2814), Fujiidera, Osaka
  - Kansai Medical University Hospital ( Site 2823), Hirakata, Osaka
  - Hamamatsu University Hospital ( Site 2874), Hamamatsu, Shizuoka
  - Matsuda Hospital ( Site 2826), Hamamatsu, Shizuoka
  - National Hospital Organization Shizuoka Medical Center ( Site 2837), Shimizu, Shizuoka
  - Institute of Science Tokyo Hospital ( Site 2827), Bunkyō, Tokyo
  - Ginza Central Clinic ( Site 2824), Chūō, Tokyo
  - The Jikei University Hospital ( Site 2843), Minato, Tokyo
  - Toranomon Hospital ( Site 2828), Minato-ku, Tokyo
  - Kitasato University Kitasato Institute Hospital ( Site 2817), Minato-ku, Tokyo
  - Kyorin University Hospital ( Site 2804), Mitaka-shi, Tokyo
  - NTT Medical Center Tokyo ( Site 2834), Shinagawa-ku, Tokyo
  - Yamanashi Prefectural Central Hospital ( Site 2836), Kofu, Yamanashi
  - Fukui Prefectural Hospital ( Site 2844), Fukui
  - Fukuoka University Hospital ( Site 2818), Fukuoka
  - Hiroshima University Hospital ( Site 2845), Hiroshima
  - Kagoshima University Hospital ( Site 2848), Kagoshima
  - Kagoshima IBD Gastroenterology Clinic ( Site 2821), Kagoshima
  - University Hospital,Kyoto Prefectural University of Medicine ( Site 2819), Kyoto
  - National Hospital Organization Kyoto Medical Center ( Site 2813), Kyoto
  - Okayama University Hospital ( Site 2870), Okayama
  - Infusion Clinic ( Site 2806), Osaka
  - National Hospital Organization Osaka National Hospital ( Site 2869), Osaka
  - Ishida Clinic of IBD and Gastroenterology ( Site 2820), Ōita
  - Saga University Hospital ( Site 2812), Saga
  - Tokitokai Tokito Clinic Coloproctology Center ( Site 2811), Saitama
  - Tokyo Yamate Medical Center ( Site 2803), Tokyo
  - Toyama Prefectural Central Hospital ( Site 2807), Toyama
  - Yamagata University Hospital ( Site 2849), Yamagata
- Latvia (3):
  - Liepaja Regional Hospital ( Site 4501), Liepāja
  - P.Stradins Clinical University Hospital Center of Gastroenterology Hepatology and Nutrition ( Site 4503), Riga
  - SIA M & M Centrs ( Site 4502), Ādaži, Ādaži
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kauno klinikos ( Site 4600), Kaunas, Kaunas County
  - VUL SANTAROS KLINIKOS ( Site 4601), Vilnius, Vilniaus Miestas
- Malaysia (4):
  - Hospital Sultanah Aminah ( Site 4702), Johor Bahru, Johor
  - Hospital Universiti Sains Malaysia ( Site 4704), Kubang Kerian, Kelantan
  - Hospital Tuanku Jaafar Seremban ( Site 4705), Seremban, Negeri Sembilan
  - Hospital Ampang ( Site 4703), Ampang, Selangor
- Mexico (9):
  - Morales Vargas Centro de Investigacion ( Site 2411), León, Guanajuato
  - PanAmerican Clinical Research - Guadalajara ( Site 2400), Guadalajara, Jalisco
  - Centro Medico Clinico Quirurgico Especializado en Investigación ( Site 2403), Tlajumulco de Zuniga, Jalisco
  - Medica Sur-Clinica de Enfermedades Digestivas y Obesidad ( Site 2406), Mexico City, Mexico City
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez" ( Site 2409), Monterrey, Nuevo León
  - Centro Multidisciplinario para el Desarrollo Especializado de la Investigacion Clinica en Yucatan ( Site 2407), Mérida, Yucatán
  - ICARO Investigaciones en Medicina ( Site 2405), Chihuahua City
  - Centro de Investigación y Gastroenterología - S.C. ( Site 2410), Mexico City
  - Oaxaca Site Management Organization S.C. ( Site 2404), Oaxaca City
- Netherlands (9):
  - Radboudumc ( Site 1402), Nijmegen, Gelderland
  - ETZ Elisabeth-Department of Gastroenterology and Hepatology ( Site 1403), Tilburg, North Brabant
  - Ziekenhuis Bernhoven-Researchbureau ( Site 1401), Uden, North Brabant
  - Onze Lieve Vrouwe Gasthuis ( Site 1405), Amsterdam, North Holland
  - Amsterdam UMC, locatie VUmc-IBD Trial Unit ( Site 1400), Amsterdam, North Holland
  - Deventer Ziekenhuis ( Site 1411), Deventer, Overijssel
  - Erasmus Medisch Centrum ( Site 1410), Rotterdam, South Holland
  - Franciscus Gasthuis & Vlietland, Locatie Gasthuis ( Site 1406), Rotterdam, South Holland
  - Universitair Medisch Centrum Utrecht ( Site 1404), Utrecht
- New Zealand (3):
  - Waikato Hospital ( Site 2903), Hamilton, Waikato Region
  - Hutt Valley District Health board HVDHB ( Site 2902), Lower Hutt, Wellington Region
  - Aotearoa Clinical Trials ( Site 2900), Auckland
- Norway (2):
  - Akershus Universitetssykehus ( Site 4200), Lørenskog, Akershus
  - Oslo Universitetssykehus Ullevål ( Site 4201), Oslo
- Poland (21):
  - Pratia Poznan ( Site 1530), Poznan, Greater Poland Voivodeship
  - Twoja Przychodnia Poznanskie Centrum Medyczne Sp. z o.o.,Twoja Przychodnia PCM ( Site 1523), Poznan, Greater Poland Voivodeship
  - Gastromed Sp. z o. o. ( Site 1513), Torun, Kuyavian-Pomeranian Voivodeship
  - Topolowa Medicenter Ryszawa & Wspolnicy sp.j. ( Site 1500), Krakow, Lesser Poland Voivodeship
  - PROMED P. LACH R. GLOWACKI SP. J. ( Site 1529), Krakow, Lesser Poland Voivodeship
  - Allmedica ( Site 1508), Nowy Targ, Lesser Poland Voivodeship
  - NZOZ FOR MED sp. z o.o. ( Site 1511), Wadowice, Lesser Poland Voivodeship
  - Planetmed ( Site 1506), Wroclaw, Lower Silesian Voivodeship
  - Vistamed & Vertigo Sp. z o.o. ( Site 1528), Wroclaw, Lower Silesian Voivodeship
  - Melita Medical ( Site 1519), Wroclaw, Lower Silesian Voivodeship
  - Penta Hospitals Przychodnie Wrocław Wejherowska ( Site 1505), Wroclaw, Lower Silesian Voivodeship
  - Centrum Zdrowia MDM ( Site 1512), Warsaw, Masovian Voivodeship
  - ETG Warszawa ( Site 1525), Warsaw, Masovian Voivodeship
  - Vivamed Sp. z o.o. ( Site 1510), Warsaw, Masovian Voivodeship
  - WIP Warsaw IBD Point Profesor Kierkuś ( Site 1503), Warsaw, Masovian Voivodeship
  - M2M Med ( Site 1526), Chorzów, Silesian Voivodeship
  - Vita Longa Sp. Zoo ( Site 1527), Katowice, Silesian Voivodeship
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne ( Site 1502), Szczecin, West Pomeranian Voivodeship
  - Sonomed Sp. z o. o. ( Site 1516), Szczecin, West Pomeranian Voivodeship
  - Med-Gastr Sp. z o.o., sp.k ( Site 1515), Lodz, Łódź Voivodeship
  - AmiCare Centrum Medyczne - Zgierska ( Site 1517), Lodz, Łódź Voivodeship
- Portugal (6):
  - Unidade Local de Saude Lisboa Ocidental - Hospital Egas Moniz ( Site 3306), Lisbon, Lisbon District
  - Unidade Local de Saude de Braga - Hospital de Braga ( Site 3300), Braga
  - Hospital dos Lusíadas Lisboa ( Site 3303), Lisbon
  - Unidade Local de Saude de Santa Maria - Hospital de Santa Maria ( Site 3305), Lisbon
  - ULSAM - Hospital de Santa Luzia ( Site 3302), Viana do Castelo
  - Unidade Local de Saude Dão-Lafões - Hospital de São Teotónio ( Site 3308), Viseu
- Romania (8):
  - MEMORIAL HEALTHCARE INTERNATIONAL S.R.L ( Site 1606), Bucharest, București
  - Monza Ares SRL ( Site 1604), Bucharest, București
  - Fundeni Clinical Institute-Gastroenterology and Hepatology Center ( Site 1608), Bucharest, București
  - Spitalul Clinic Judetean de Urgenta Cluj Napoca-Gastroenterology ( Site 1605), Cluj-Napoca, Cluj
  - GastroMed ( Site 1609), Cluj-Napoca, Cluj
  - Spitalul Clinic Judetean Mures-Gastroenterology ( Site 1607), Târgu Mureş, Mureș County
  - S.C Centrul de Gastroenterologie Dr. Goldis S.R.L-Gastroenterology ( Site 1601), Timișoara, Timiș County
  - Asociatia Oncohelp ( Site 1610), Timișoara, Timiș County
- Serbia (5):
  - Clinical Hospital Center Dragisa Misovic ( Site 1708), Belgrade, Beograd
  - Clinical Hospital Center Zvezdara-Gastroenterology and hepatology Department ( Site 1705), Belgrade, Beograd
  - University Medical Center "Bezanijska kosa"-Gastroenterology and hepatology ( Site 1704), Belgrade, Beograd
  - Clinical Center Kragujevac ( Site 1703), Kragujevac, Beograd
  - General Hospital "Djordje Joanovic" ( Site 1707), Zrenjanin, Srednjebanatski Okrug
- Singapore (2):
  - Singapore General Hospital ( Site 4801), Singapore, Central Singapore
  - Tan Tock Seng Hospital-Gastroenterology and Hepatology ( Site 4800), Singapore, Central Singapore
- Slovakia (8):
  - Breznianske centrum gastroenterologie ( Site 1806), Brezno, Banská Bystrica Region
  - Fakultna nemocnica s poliklinikou F.D.Roosevelta Banska Bystrica ( Site 1802), Slovakia, Banská Bystrica Region
  - Cliniq s.r.o. ( Site 1800), Bratislava, Bratislava Region
  - ENDOMED ( Site 1801), Košice, Košice Region
  - KM Management ( Site 1804), Nitra, Nitra Region
  - Accout Center ( Site 1805), Šahy, Nitra Region
  - GASTRO I ( Site 1807), Prešov, Presov
  - Gastro LM ( Site 1808), Prešov, Presov
- South Africa (6):
  - Wits Clinical Research-Research ( Site 3208), Johannesburg, Gauteng
  - Wits Clinical Research-Wits Clinical Research Bara ( Site 3206), Soweto, Gauteng
  - Panorama Medical Centre ( Site 3209), Cape Town, Western Cape
  - Spoke Research ( Site 3210), Cape Town, Western Cape
  - Life Kingsbury Hospital ( Site 3203), Cape Town, Western Cape
  - Private Practice - Dr. M.N. Rajabally ( Site 3213), Cape Town, Western Cape
- South Korea (14):
  - Wonju Severance Christian Hospital-Internal Medicine ( Site 3003), Wŏnju, Kang-won-do
  - The Catholic University Of Korea St. Vincent's Hospital-Gastroenterology ( Site 3006), Suwon, Kyonggi-do
  - Dong-A University Hospital ( Site 3010), Busan, Pusan-Kwangyokshi
  - Inje University Haeundae Paik Hospital ( Site 3009), Haeundae-gu, Pusan-Kwangyokshi
  - Chung-Ang University Hospital ( Site 3008), Dongjak-gu, Seoul
  - Yeungnam University Medical Center ( Site 3004), Daegu, Taegu-Kwangyokshi
  - The Catholic University of Korea, Daejeon St. Mary's Hospital ( Site 3011), Daejeon, Taejon-Kwangyokshi
  - Kyung Hee University Hospital ( Site 3013), Seoul
  - Seoul National University Hospital ( Site 3005), Seoul
  - Kangbuk Samsung Hospital-Internal Medicine ( Site 3002), Seoul
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital ( Site 3012), Seoul
  - Severance Hospital, Yonsei University Health System-Department of Internal Medicine ( Site 3000), Seoul
  - Asan Medical Center ( Site 3007), Seoul
  - Samsung Medical Center ( Site 3001), Seoul
- Spain (11):
  - Hospital Germans Trias i Pujol ( Site 3413), Badalona, Barcelona
  - Hospital Universitari Mutua Terrassa ( Site 3416), Terrassa, Barcelona
  - Hospital Galdakao-Usansolo ( Site 3409), Galdakao-Usansolo, Bizkaia
  - Hospital Universitario de Fuenlabrada-Digestive ( Site 3415), Fuenlabrada, Madrid
  - Hospital La Princesa-Gastroenterology ( Site 3411), Madrid, Madrid, Comunidad de
  - Fundación Jimenez Diaz ( Site 3420), Madrid, Madrid, Comunidad de
  - Hospital Universitario de Torrejon ( Site 3417), Torrejón de Ardoz, Madrid, Comunidad de
  - Hospital Universitari i Politecnic La Fe-Enfermedad Inflamatoria Intestinal ( Site 3405), Valencia, Valencia
  - HOSPITAL CLINICO DE VALENCIA ( Site 3406), Valencia, Valenciana, Comunitat
  - HOSPITAL GENERAL UNIVERSITARIO GREGORIO MARAÑON-Aparato Digestivo ( Site 3403), Madrid
  - Hospital Universitario La Paz-Unidad de Enfermedad Inflamatoria Intestinal ( Site 3402), Madrid
- Sweden (4):
  - Danderyds Sjukhus ( Site 4401), Danderyd, Stockholm County
  - Karolinska Universitetssjukhuset Solna ( Site 4400), Stockholm, Stockholm County
  - Akademiska Sjukhuset ( Site 4403), Uppsala, Uppsala County
  - Universitetssjukhuset i Linköping ( Site 4402), Linköping, Östergötland County
- Switzerland (3):
  - INTESTO-Gastroenterologische Praxis / Crohn-Colitis Zentrum Bern ( Site 1902), Bern, Canton of Bern
  - Cantonal Hospital St.Gallen-Klinik für Gastroenterologie / Hepatologie ( Site 1901), Sankt Gallen, Canton of St. Gallen
  - UniversitätsSpital Zürich-Gastroenterologie & Hepatologie ( Site 1900), Zurich, Canton of Zurich
- Taiwan (5):
  - Changhua Christian Hospital ( Site 3104), Changhua County, Changhua
  - National Taiwan University BioMedical Park Hospital ( Site 3103), Zhubei, Hsinchu
  - China Medical University Hospital ( Site 3100), Taichung
  - National Taiwan University Hospital ( Site 3102), Taipei
  - Chang Gung Medical Foundation-Linkou Branch ( Site 3101), Taoyuan District
- Turkey (Türkiye) (9):
  - Istanbul Universitesi Cerrahpasa-Internal Diseases ( Site 3503), Istanbul- Fatih, Istanbul
  - ANKARA UNIVERSITY IBNI SINA HOSPITAL ( Site 3507), Ankara
  - Hacettepe Universite Hastaneleri ( Site 3500), Ankara
  - Ankara Bilkent Şehir Hastanesi-Gastroenterology ( Site 3501), Ankara
  - Antalya Egitim ve Arastirma Hastanesi ( Site 3508), Antalya
  - Trakya University Medical Faculty Hospital ( Site 3510), Edirne
  - Eskisehir Osmangazi University Faculty of Medicine ( Site 3512), Eskişehir
  - Marmara Universitesi Pendik Egitim Arastirma Hastanesi ( Site 3505), Istanbul
  - Kocaeli University Medical Faculty Hospital ( Site 3509), Kocaeli
- Ukraine (10):
  - Communal non-profit enterprise "Regional clinical hospital of Ivano-Frankivsk Regional Council" ( Site 4115), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Center of Family Medicine Plus-Treatment Prevention Unit ( Site 4103), Kyiv, Kyivska Oblast
  - Communal Non-profit Enterprise of Lviv Regional Council "Lviv Regional Clinical Hospital"-proctology ( Site 4109), Lviv, Lviv Oblast
  - Limited liability company "Medical center Health Clinic"-Gastroenterology, Hepatology and Endocrino ( Site 4107), Vinnytsia, Vinnytsia Oblast
  - Municipal Nonprofit Enterprise "Vinnytsia Regional Clinical -Gastroenterology department ( Site 4114), Vinnytsia, Vinnytsia Oblast
  - Communal Non-Commercial Enterprise "Vinnytsia City Clinical -Clinical Therapeutic Department #1 ( Site 4111), Vinnytsia, Vinnytsia Oblast
  - Municipal Enterprise "Volyn Regional Clinical Hospital" of V-surgery department (abdominal, colopro ( Site 4113), Lutsk, Volyn Oblast
  - Medical Center "Universal Clinic "Oberig" of Limited Liability Company "Kapytal" ( Site 4100), Kyiv
  - Dobrobut Medical Center ( Site 4101), Kyiv
  - Medical Center of Private Enterprise "Sygma" ( Site 4108), Kyiv
- United Kingdom (10):
  - Southmead Hospital ( Site 2004), Bristol, Bristol, City of
  - Addenbrooke's Hospital ( Site 2005), Cambridge, Cambridgeshire
  - Royal Devon & Exeter Hospital-IBD Research Group ( Site 2001), Exeter, Devon
  - Doncaster Royal Infirmary ( Site 2006), Doncaster, England
  - Huddersfield Royal Infirmary ( Site 2010), Huddersfield, England
  - Whipps Cross University Hospital-Clinical Research Unit ( Site 2000), London, England
  - St. George's Hospital ( Site 2007), London, England
  - Southampton General Hospital-Gastroenterology ( Site 2003), Southampton, Hampshire
  - University College London Hospital-Clinical Research Facility ( Site 2002), London, London, City of
  - Walsall Manor Hospital ( Site 2009), West Midlands, Walsall

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26193&tenant=MT_MSD_9011